CLINICAL TRIAL: NCT06349109
Title: Physical Activity Level and Determinants in Children With Wolff-Parkinson-White Syndrome
Brief Title: Physical Activity in Children With Wolff-Parkinson-White Syndrome
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Haluk Tekerlek, Research assistant, PhD, Karamanoğlu Mehmetbey University
Other Study IDs: PA-WPW
Record Dates: First submitted 2024-03-30; First posted 2024-04-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Wolff-Parkinson-White Syndrome
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WPW group
  Interventions: Other: Cardiopulmonary exercise test; Other: Atrial-Ventricular Strain Analysis; Other: Arterial Stiffness Measurement; Other: Physical Activity Level; Other: Physical Activity Barriers Assesment
- Control Group
  Interventions: Other: Physical Activity Level; Other: Physical Activity Barriers Assesment

INTERVENTIONS:
Other: Cardiopulmonary exercise test — The cardiopulmonary exercise test (CPET), the gold standard for the assessment of cardiorespiratory fitness, will be used. The Modified Bruce/half Bruce protocol with will be used. In addition, dyspnoea, leg fatigue and general fatigue will be recorded every three minutes at rest, during the test and during the post-test recovery phases using the Modified Borg Scale and blood pressure will be recorded with a sphygmomanometer. The test will be continued until individuals reach the end of the protocol or until the last point at which they wish to stop the test. The test will be terminated if the patient wishes to terminate the test, severe breathlessness, leg fatigue or general fatigue, loss of coordination, progressive chest pain, ST segment elevation or depression of more than 2 mm, oxygen saturation of 80% or less, reaching 85% or more of the predicted heart rate. Oxygen consumption (VO2peak) will be used as the primary outcome measure for cardiorespiratory fitness.
  Groups: WPW group
Other: Atrial-Ventricular Strain Analysis — Atrial-Ventricular strain will be evaluated by a specialist physician using Speckle Tracking Echocardiography. During the evaluation, standard echocardiographic measurements will be made with transthoracic echocardiography. With these measurements, images suitable for strain analysis will be obtained. Deformation analysis will be performed using the speckle tracing method for the appropriate images obtained and hemodynamic parameters obtained by the analysis will be recorded.
  Groups: WPW group
Other: Arterial Stiffness Measurement — Arterial stiffness will be assessed using the pulse wave velocity (PWV) technique with the Mobile-O-GRAPH (TG) (LE.M., Stolberg, Germany), an oscillometer-based device. After the patients have rested sufficiently, measurements will be taken in an upright sitting position in a quiet and sufficiently bright environment at room temperature, with the device manso placed 2-3 cm above the chiibital fossa in the non-dominant upper limb and the arms raised to the level of the heart. Pulse propagation velocity will be calculated in m/sec with the help of a computer. A high velocity data indicates a high level of arterial stiffening and a low velocity data indicates a low level of arterial stiffening.
  Groups: WPW group
Other: Physical Activity Level — Physical activity level will be assessed with the Child Physical Activity Questionnaire.
Other: Physical Activity Barriers Assesment — "Physical Activity Outcome Expectancies (child survey)" and "Physical Activity Home Environment Scale (Child)" will be used in children, while " Physical activity barriers (Parent)" will be used in family members.

SUMMARY:
The aim of this study was to investigate the level of physical activity and its determinants in children with WPW.

ELIGIBILITY:
Inclusion Criteria:

* Being between 7-18 years old
* Ensuring clinical stability in patients
* No change in drug therapy, if any, that adversely affects clinical stability

Exclusion Criteria:

* Neurological and/or genetic musculoskeletal disorders
* Diagnosed orthopaedic and cognitive problems that prevent the tests from being performed
* History before 4 weeks of cardiac or other body system problems
* The patient and/or his/her family does not want to be included in the study

Ages: 7 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients aged 7-18 years who are followed up by the Department of Paediatrics, Division of Paediatric Cardiology, Faculty of Medicine of a university will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The Physical Activity Questionnaire for Older Children Score | 15-20 mins
  The PAQ-C comprises ten items and higher scores indicate a higher level of activity. The first item of the PAQ-C consists of 22 common sports and leisure activities for which the participants select the score based on the frequency of the activity performed during the preceding seven days on a five-point rating scale, after which a mean composite score was calculated. The remaining eight items address physical activities performed during the day, for example, physical education classes, recess time, lunchtime, as well as afterschool activities on weekday evenings and weekends, and finally a summary for all days of the week. The mean score of the first nine items is the summary score of the PAQ-C. The tenth item inquires about any unusual circumstances (e.g., sickness) that affected/prevented the child's physical activity in the seven days preceding the assessment.

SECONDARY OUTCOMES:
VO2peak | 30-45 minutes
  Peak oxygen uptake
aPWV | 15-20 minutes
  Arterial pulse wave velocity
GLS | 30-45 minutes
  Global longitudinal strain for LV function
LASr | 30-45 minutes
  Left atrial strain - Reservuar
LASct | 30-45 minutes
  Left atrial strain - Contractile
LAScd | 30-45 minutes
  Left atrial strain - Conduit
Physical activity barriers (Parent) scale score | 15-20 minutes
  The original scale consists of 13 items and two dimensions. The Turkish adapted version of the scale consists of two dimensions and 11 items. Items 1-6 in the scale constitute the "Environmental barriers" sub-dimension and items 7-11 constitute the "Personal barriers" sub-dimension. Total scores are obtained separately for the two sub-dimensions of the scale. The score range varies between 6 (min) and 30 (max) for the "Environmental barriers" sub-dimension and between 5 (min) and 25 (max) for the "Personal barriers" sub-dimension. The higher score in the sub-dimensions indicates the magnitude of the barriers to physical activity in those areas for the participant.
Physical Activity Outcome Expectancies (Child) scale score | 15-20 minutes
  The scale is a three-point Likert-type scale consisting of 17 items and two dimensions. The "Negative outcome expectancies" sub-dimension of the scale consists of items 2, 3, 4, 6, 7, 11, 12, 14 and 16 and the "Positive outcome expectancies" sub-dimension consists of items 1, 5, 8, 9, 10, 13, 15 and 17. Total scores are obtained separately for the two dimensions. The score that can be obtained from the 9 items related to the negative outcome expectancies sub-dimension varies between 9 and 17. The score that can be obtained from 8 items related to the positive outcome expectancy sub-dimension varies between 8 and 24. A high score in the negative outcome expentancies sub-dimension indicates an excess of negative expectations about physical activity. A high score on the Positive Outcome Expentancies sub-dimension indicates an excess of positive expectations about physical activity.
Physical Activity Home Environment (Child) scale score | 15-20 minutes
  The scale is a triple likert type scale consisting of 5 items. - The score range of the scale is 5-15. - A high score on the scale indicates that the family supports the child to be more physically active.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No